CLINICAL TRIAL: NCT01516398
Title: Endothelin-1 (ET-1) Levels as Predictors of Pulmonary Hypertension Risk in Premature Infants With Bronchopulmonary Dysplasia (BPD)
Brief Title: Predictors of Pulmonary Hypertension Risk in Premature Infants With Bronchopulmonary Dysplasia
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Christine Johnson, Principle Investigator, Stanford University
Other Study IDs: BPD22044
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Bronchopulmonary Dysplasia (BPD); Hypertension, Pulmonary
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Preterm infants: No interventions were performed. Group consisted of preterm infants enrolled in the study.
- Term control infants: No interventions were performed. Group consisted of term infants enrolled in the study to serve as controls for the preterm infant group.

SUMMARY:
A lung condition called bronchopulmonary dysplasia (BPD) is a major cause of poor outcomes and death for premature infants. Infants with BPD are also at high risk for pulmonary hypertension (PH)-an important contributor to their condition. Previous research has suggested that a protein in the blood, endothelin-1 (ET-1), is associated with pulmonary disease.

This study aims to investigate the incidence of PH and levels of ET-1 among premature babies with BPD. It will also potentially allow us to focus further research efforts and treatment towards these infants, some of our sickest patients at LPCH.

DETAILED DESCRIPTION:
This study aims to 1) investigate the incidence of PH among premature infants with BPD versus those without BPD and 2) investigate ET-1 levels in infants with BPD-associated PH versus those without BPD-associated PH. This study will allow us to help define a high-risk population at LPCH-namely, premature infants with BPD-associated PH. It will also potentially allow us to focus further research efforts and treatment targets towards these infants who encompass some of our sickest patients at LPCH.

In 2009 the Division of Lung Diseases of the National Heart, Lung and Blood Institute (NHLBI) published seven priority areas for research in pediatric pulmonary diseases, one of which was pulmonary vascular disease. An emphasis was made on finding 'clinical strategies that anticipate the development of PH [which] may allow earlier recognition and more aggressive therapy, thereby slowing the development of PH in many chronic lung parenchymal and vascular diseases'. This study attempts to address this goal. Specifically we aim to evaluate ET-1 levels in premature infants diagnosed with BPD and with BPD-associated PH. If ET-1 levels are found to correlate with disease state the possibility of prediction and possible early treatment for PH in these infants is raised and merits investigation.

ELIGIBILITY:
Inclusion Criteria:

* Premature Infants (<30 weeks EGA)

Exclusion Criteria:

* Major congenital malformations (cardiac, respiratory, gastrointestinal)
* congenital infection, and/or
* known genetic syndromes (i.e. trisomy 21)

Max Age: 30 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: LPCH premature neonates
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
Infant develops BPD | 36 weeks of age

SECONDARY OUTCOMES:
Infant develops PH | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christine Johnson, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - El Camino Hospital, Mountain View, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California

IPD SHARING:
Plan to Share IPD: Yes
Publication